CLINICAL TRIAL: NCT05643079
Title: Medial Displacement Calcaneal Osteotomy and FDL- Transfer - a Prospective Comparative Study Between Metal/Bio-Tenodesis Screw (Arthrex) and the Human, Allogeneic Cortical Bone Screw (Shark Screw®️, Surgebright-GmbH)
Brief Title: Medial Displacement Calcaneal Osteotomy and FDL- Transfer - With a Human, Allogeneic Cortical Bone Screw
Status: Recruiting | Type: Observational
Sponsor: Orthopedic Hospital Vienna Speising (Other)
Responsible Party: Principal Investigator, Forian Wenzel-Schwarz, Senior Physician Dr. med., Orthopedic Hospital Vienna Speising
Other Study IDs: FDLTransferSharkScrew
Record Dates: First submitted 2022-10-21; First posted 2022-12-08 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Flat Feet; Flexor Tendon Rupture; Tibialis Posterior Dysfunction; Deformity, Foot
Keywords: human allogeneic cortical bone screw; Shark Screw®; flat foot deformity; FDL Transfer; Tibialis posterior dysfunction; metal screw; Bio-Tenodesis screw; flat foot
MeSH Terms: conditions — Flatfoot; Posterior Tibial Tendon Dysfunction; Foot Deformities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- metal/Bio-Tenodesis group: medializing calcaneal osteotomy, debridement of the tibialis posterior tendon, and/or transfer of the flexor digitorum longus (FDL) tendon with the following screws:
  Metal-/Bio-Tenodesis screw (Arthrex, Naples, Florida, USA)
  Metal-Screw:
  ø 6,7 mm length: 40-60 mm
  Bio-Tenodesis screw:
  ø 4,00 mm, length: 10 mm ø 4,75 mm, length: 15 mm ø 5,50 mm, length: 15 mm
  Interventions: Procedure: medializing calcaneal osteotomy and/or transfer of the flexor digitorum longus tendon (FDL) with metal/Bio-Tenodesis screws
- human, allogeneic cortical bone screw (Shark Screw®): medializing calcaneal osteotomy, debridement of the tibialis posterior tendon, and/or transfer of the flexor digitorum longus (FDL) tendon with the following screws:
  Shark Screw® (Surgebright-GmbH, 4040 Lichtenberg, Austria)
  Versions used:
  Shark Screw® diver ø: 5,0 mm, length: 35 mm Shark Screw® diver ø: 5,0 mm, length: 45 mm Shark Screw® tendon ø: 5,0 mm, length: 15 mm
  Interventions: Procedure: medializing calcaneal osteotomy and/or transfer of the flexor digitorum longus tendon (FDL) with Shark Screws®

INTERVENTIONS:
Procedure: medializing calcaneal osteotomy and/or transfer of the flexor digitorum longus tendon (FDL) with metal/Bio-Tenodesis screws — The calcaneus osteotomy is performed dorsal proximal to plantar distal with caution of the peroneal tendons and sural nerve. After mobilization the dorsal fragment is displaced medially by~10mm. Thereafter, a guide wire is placed from plantar-lateral into the ventral portion of the calcaneus under fluoroscopic control. After stab incision and length measurement, the osteotomy is fixed with a Metal/Bio-Tenodesis screw(MBS). The lateral projection of the edge is straightened. Opening of the tendon sheath of the FDL muscle and dissection distally to Henry's node. Settling of the tendon and arming with a "shuttle suture". Tendon diameter measurement. Place a guide wire at os naviculare directed from plantar to dorsal in 20°proximal guidance. Pull through the FDL tendon from plantar to dorsal and fixation with an MBS in 20°of pointed foot position and inversion with appropriate desired tension. The tendon is then sutured to the stump of the tibialis posterior tendon, retinaculum sutures.
  Other Names: Metal/Bio-Tenodesis screw intervention
  Groups: metal/Bio-Tenodesis group
Procedure: medializing calcaneal osteotomy and/or transfer of the flexor digitorum longus tendon (FDL) with Shark Screws® — The calcaneus osteotomy is performed dorsal proximal to plantar distal with caution of the peroneal tendons and sural nerve. After mobilization the dorsal fragment is displaced medially by approx.10mm. Thereafter, a guide wire is placed from plantar-lateral into the ventral portion of the calcaneus under fluoroscopic control. After stab incision and length measurement, the osteotomy is fixed with a Shark Screw®. The lateral projection of the edge is straightened. Opening of the tendon sheath of the FDL muscle and dissection distally to Henry's node. Settling of the tendon and arming with a "shuttle suture". Tendon diameter measurement. Place a guide wire at os naviculare directed from plantar to dorsal in 20°proximal guidance. Pull through the FDL tendon from plantar to dorsal and fixation with the Shark Screw® in 20°of pointed foot position and inversion with appropriate desired tension. The tendon is then sutured to the stump of the tibialis posterior tendon, retinaculum sutures.
  Other Names: Shark Screw® intervention
  Groups: human, allogeneic cortical bone screw (Shark Screw®)

SUMMARY:
The goal of this observational study is to compare the use of a screw made of human bone (Shark-Screw®, Surgebright-GmbH) with the metal/Bio-Tenodesis screw (Arthrex) in the treatment of the symptomatic flatfoot using the medializing calcaneus osteotomy with flexor digitorum longus transfer (FDL) in adult patients. The advantage of the human bone screw is that after surgery no hardware removal is necessary. The screw is transformed from the body to normal bone.

The main questions it aims to answer are:

* Can the human bone screw achieve union rates like the metal/Bio-Tenodesis screw?
* Is the time to union similar between the different screws?
* Is the complication rate similar between the different screws?
* Are the activity scores American Orthopaedic Foot and Ankle Society (AOFAS), Foot and Ankle Outcome Score (FAOS) and Foot Function Index (FFI) after surgery similar in the compared patient groups?

Participants will have

* the surgery
* follow-ups at 6 weeks, 6 months, 1 and 2 years.
* X-rays are performed at each follow up.
* CT-scans are performed after 6 months.
* activity scores are collected at the follow up after 6 months, 1 year and 2 years.

DETAILED DESCRIPTION:
Symptomatic flatfoot deformity in adults often occurs as a result of dysfunction of the Tibialis posterior tendon (TPTD), with a prevalence of 3.3%. Structured non-surgical treatment programs with orthotics and physiotherapy can achieve a high level of long-term subjective and functional satisfaction, with surgery being avoided in 70-89% of cases. Surgical intervention is indicated for progressive or uncontrolled symptoms. Flexible flatfoot deformity, stage II classified by Johnson and Strom, can be treated with a joint-preserving strategy, which usually includes a medializing calcaneal osteotomy, debridement of the tibialis posterior tendon, and transfer of the flexor digitorum longus (FDL) tendon. 87% satisfaction after ten years was observed in both pain relief and foot function and alignment.

Metal screws have been used for decades to treat bone fractures. The removal is the major disadvantage of conventional osteosyntheses and requires a second operation, with all the resulting risks of complications for each patient. The use of the bone screw from allogeneic cortical bone would reduce costs substantially, with a significant reduction in the average complication rate to 0.3%.

The idea of stabilizing fractures using compact bone instead of metal is not new. Obwegeser published the clinical use of 796 screw implants of allogeneic bone and reported that the only complication was the fracture of 6 screws (<1%) and three screw loosening (<0,5%).

Since 2016, the human, allogeneic cortical bone screw(Shark Screw®) has been used by two tissue banks, the Austrian Austrian tissue bank Surgebright-GmbH and the German Institute for Cell and Tissue Replacement (DIZG). The Shark Screw® graft was approved by the competent Austrian authority (AGES) in 2016. The bone graft immediately creates a solid, purely bony connection. This leads to bone remodeling, bone incorporation and optimal reparation in the surgical area. Depending on the loads and requirements, the bone connection adapts for the future. The bone grafts undergo a certified sterilization procedure at the DIZG, which was developed in 1985 at the Berlin Charité.

Due to the lack of further systematic investigations to objectively confirm the theoretically given and subjectively experienced product advantages, this observational study is now being conducted.

The aim of the present study is to evaluate the application of the human allogeneic cortical bone screw (Shark Screw®) and the metal/Bio-Tenodesis screw in the surgical treatment (medializing calcaneus osteotomy with FDL transfer) of symptomatic flatfoot and to systematically document corresponding clinical and radiological parameters before and after surgery.

ELIGIBILITY:
Inclusion Criteria

* Indication for the use of a metal/Bio-Tenodesis screw or human bone screw in medializing calcaneus osteotomy with FDL transfer.
* BMI< 40 kg/m²

Exclusion Criteria:

* Insufficient knowledge of German
* Alcohol and drug abuse
* Pregnant woman or nursing mother
* Foreseeable compliance problems
* Neoplastic diseases, malignant bone tumors, rheumatoid arthritis
* Active osteomyelitis
* History of foot surgery
* Advanced osteoarthritis of the lower ankle joint
* Ulcerations in the skin of the surgical area
* Immunosuppressive medications that cannot be discontinued
* BMI >40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with an indication for the use of a metal/Bio-Tenodesis screw or human bone screw in medializing calcaneus osteotomy with/without FDL transfer.
  The patient has the choice of the treatment method after explanation advantages and disadvantages for each surgery method
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
x-ray qualitative evaluation of changes in bony union of calcaneus osteotomy | 6 weeks, 6 months, 1 year, 2 years
  bony union will be evaluated
CT-scan qualitative evaluation of changes in bony union of calcaneus osteotomy | 6 months, 1 year
  bony union will be evaluated

SECONDARY OUTCOMES:
changes in AOFAS score in comparison to presurgery | 6 months, 1 year and 2 years
  The American Orthopedic Foot and Ankle Score (AOFAS) units in percent (%), the higher the better
changes in Foot and Ankle Outcome Score (FOAS) score in comparison to presurgery | 6 months, 1 year and 2 years
  Foot and Ankle Outcome Score units in percent (%), the higher the better
changes in FFI score in comparison to presurgery | 6 months, 1 year and 2 years
  Foot Function Index units in percent (%), the higher the better
changes in Vas-Pain score in comparison to presurgery | 6 weeks, 6 months, 1 year and 2 years
  Visual Analog Scale Pain Score values between 0 and 10, 0= no pain, 10 sever pain
complications | during surgery, 6 weeks, 6 months, 1 year and 2 years
  Complications will be recorded during surgery and the kind of complication described, number of patients with complications are given
reoperations | during surgery, 6 weeks, 6 months, 1 year and 2 years
  Reoperations will be recorded when needed and the kind of re-operation and number of patients with reoperations are given
pseudoarthrosis | during surgery, 6 months, 1 year and 2 years
  Pseudarthrosis will be recorded at the follow up at 2 years and number of patients with Pseudarthrosis are given

CONTACTS AND LOCATIONS:
Overall Officials: Florian Wenzel-Schwarz, MD, Principal Investigator — Abteilung für Kinderorthopädie und Fußchirurgie Orthopädisches Spital Speising, Vienna, Austria
Locations (1):
- Abteilung für Kinderorthopädie und Fußchirurgie Orthopädisches Spital Speising, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
due to the sensibility of the row data individual data will only be available on request

REFERENCES:
- [Background] Pastl K, Pastl E, Flory D, Borchert GH, Chraim M. Arthrodesis and Defect Bridging of the Upper Ankle Joint with Allograft Bone Chips and Allograft Cortical Bone Screws (Shark Screw(R)) after Removal of the Salto-Prosthesis in a Multimorbidity Patient: A Case Report. Life (Basel). 2022 Jul 11;12(7):1028. doi: 10.3390/life12071028. PMID 35888116
- [Background] Pastl K, Schimetta W. The application of an allogeneic bone screw for osteosynthesis in hand and foot surgery: a case series. Arch Orthop Trauma Surg. 2022 Oct;142(10):2567-2575. doi: 10.1007/s00402-021-03880-6. Epub 2021 Apr 8. PMID 33834287
- [Background] Brcic I, Pastl K, Plank H, Igrec J, Schanda JE, Pastl E, Werner M. Incorporation of an Allogenic Cortical Bone Graft Following Arthrodesis of the First Metatarsophalangeal Joint in a Patient with Hallux Rigidus. Life (Basel). 2021 May 24;11(6):473. doi: 10.3390/life11060473. PMID 34073841
- [Background] Johnson KA, Strom DE. Tibialis posterior tendon dysfunction. Clin Orthop Relat Res. 1989 Feb;(239):196-206. PMID 2912622
- [Background] Obwegeser JA. [Absorbable and bioconvertible osteosynthesis materials in maxillofacial surgery]. Mund Kiefer Gesichtschir. 1998 Nov;2(6):288-308. doi: 10.1007/s100060050077. German. PMID 9880999
- [Background] Hanslik-Schnabel B, Flory D, Borchert GH, Schanda JE. Clinical and Radiologic Outcome of First Metatarsophalangeal Joint Arthrodesis Using a Human Allogeneic Cortical Bone Screw. Foot Ankle Orthop. 2022 Jul 29;7(3):24730114221112944. doi: 10.1177/24730114221112944. eCollection 2022 Jul. PMID 35924004
- [Background] Amann P, Pastl K, Neunteufel E, Bock P. Clinical and Radiologic Results of a Human Bone Graft Screw in Tarsometatarsal II/+III Arthrodesis. Foot Ankle Int. 2022 Jul;43(7):913-922. doi: 10.1177/10711007221081533. Epub 2022 Apr 2. PMID 35373594
- [Background] Sailer S, Lechner S, Flossmann A, Wanzel M, Habeler K, Krasny C, Borchert GH. Treatment of scaphoid fractures and pseudarthroses with the human allogeneic cortical bone screw. A multicentric retrospective study. J Orthop Traumatol. 2023 Feb 10;24(1):6. doi: 10.1186/s10195-023-00686-7. PMID 36765020
- [Background] Krasny C, Radda C, Polke R, Schallmayer D, Borchert GH, Albrecht C. A human, allogeneic cortical bone screw for distal interphalangeal joint (DIP) arthrodesis: a retrospective cohort study with at least 10 months follow-up. Arch Orthop Trauma Surg. 2023 Jul;143(7):4557-4564. doi: 10.1007/s00402-023-04785-2. Epub 2023 Feb 9. PMID 36757467